CLINICAL TRIAL: NCT02764060
Title: The Effect of Tongue Scraping Compared to Tongue Cleaning on the Tongue Coating of Periodontitis Patients
Brief Title: The Effect of Tongue Cleaning in Periodontitis Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s54161
Record Dates: First submitted 2016-04-27; First posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-04

CONDITIONS: Periodontitis; Tongue Coating
Keywords: Periodontitis; Tongue coating; Tongue cleaning; Bacterial load
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tongue scraper (Experimental): In this group the subjects are explained how to use a plastic loop-formed tongue cleaner (Halita® tongue cleaner (Dentaid, Spain)) to clean their tongues.
  Interventions: Device: Tongue scraper
- Toothbrush (Experimental): In this group the subjects are explained how to use a toothbrush (Oral-B® Indicator® medium tooth brush) to clean their tongues.
  Interventions: Device: Toothbrush

INTERVENTIONS:
Device: Tongue scraper — The patients were instructed to start cleaning the tongue by two pulling strokes along the median sulcus of the tongue, followed by two pulling strokes along the lateral edges of the tongue.
  Other Names: Tongue scraper (Halita® tongue cleaner (Dentaid, Spain))
  Arms: Tongue scraper
Device: Toothbrush — The patients who were assigned to the tooth brush group were taught to perform three forward and backward strokes along the median sulcus and at each lateral part of the tongue.
  Other Names: Toothbrush (Oral-B® Indicator® medium tooth brush)
  Arms: Toothbrush

SUMMARY:
The aim of this study was to examine in periodontitis patients with visible tongue coating the changes in microbial load (aerobic and anaerobic) of the 14 day use of a tongue scraper versus the use of a regular toothbrush to clean the tongue.

DETAILED DESCRIPTION:
Volatile sulphur compounds (VSC's) are the most important causes of bad breath. Since the micro-organisms that produce VSC's are also periodopathogens, intuitively, one would think that there is a positive correlation between VSC levels in exhaled breath and periodontitis. However, not all periodontitis patients have bad breath. A possible explanation can be a positive relationship between tongue coating an bad breath. In the past, tongue cleaning was already researched in an oral healthy population. This research aimed to examine in periodontitis patients with visible tongue coating the changes in microbial load (aerobic and anaerobic) of the 14 day use of a tongue scraper versus the use of a regular toothbrush to clean the tongue. Additionally changes in tongue coating; and patient perception about tongue cleaning was researched.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy patients
* periodontitis patients

Exclusion Criteria:

* already using a tongue cleaning device
* use of antibiotics the previous 6 months
* rinsing with a chlorhexidine mouth rinse the past month
* smokers
* patients who underwent periodontal therapy the past three years were not included.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Extension of the tongue coating | 14 days
  Extension of the tongue coating measured according to Miyazaki (1995) and Winkel (2003).

SECONDARY OUTCOMES:
Bacterial load measured by culturing methods | 14 days
  Microbiological composition of the tongue coating.
Bacterial load measured by means of qPCR | 14 days
  Microbiological composition of the tongue coating.
Bacterial composition of unstimulated saliva (measured with the aid of culturing methods) | 14 days
  Microbiological composition of the saliva.
Bacterial composition of unstimulated saliva (measured with qPCR) | 14 days
  Microbiological composition of the saliva.
Experience of the subject of tongue coating related factors measured using a questionnaire | 14 days
  Experience of the subject of the breath odour, taste perception; and cleanliness of the tongue.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Quirynen, Study Director — marc.quirynen@uzleuven.be
Locations (1):
- UZLeuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quirynen M, Avontroodt P, Soers C, Zhao H, Pauwels M, van Steenberghe D. Impact of tongue cleansers on microbial load and taste. J Clin Periodontol. 2004 Jul;31(7):506-10. doi: 10.1111/j.0303-6979.2004.00507.x. PMID 15191584